CLINICAL TRIAL: NCT07168044
Title: A Community Cardiovascular Disease Risk Reduction Program in Older Adults Engaged in Congregate Nutrition Services (CAN-DO)
Acronym: Can-Do
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Martha Biddle (Other)
Responsible Party: Sponsor-Investigator, Martha Biddle, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 103470; 1013170404 (Other Grant/Funding Number: University of Kentucky College of Nursing)
Record Dates: First submitted 2025-08-05; First posted 2025-09-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Risk Reduction; Cardiovascular Risk
Keywords: Community health worker; cardiovascular risk reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAN DO (Experimental): usual programing offered as part of the congregate meal program plus 18 weekly group education sessions related to CVD risk reduction and nutrition.
  Interventions: Behavioral: CAN-DO

INTERVENTIONS:
Behavioral: CAN-DO — usual programing offered as part of the congregate meal program plus 18 weekly group education sessions related to CVD risk reduction and nutrition.

SUMMARY:
Investigators plan to test the effect of a Cardiovascular disease (CVD) risk reduction program targeted to improve nutrition and self-management of chronic cardiovascular conditions among older adults participating in congregate meal programs offered at community senior centers.

DETAILED DESCRIPTION:
This project proposes utilizing community health workers (CHWs) to deliver targeted health programming to participants in congregate meal programs as part of the Title III-C Nutrition Services Program. By integrating a targeted intervention into these community settings, this proposal aims to enhance individual health outcomes and support healthy nutrition among older adults. This approach prioritizes an evidence based, responsive, community-based solution to the increasingly complex health needs of this expanding population, fostering healthier aging and more resilient communities.

The purpose of this study is to examine the feasibility of a CVD risk reduction program targeted to improve nutrition and self-management of chronic cardiovascular conditions among older adults participating in congregate meal programs offered at community senior centers. The specific aim is to examine the feasibility of a CVD risk reduction program (CAN-DO) delivered to older adults participating in a congregate meal program. The rates of recruitment, retention, acceptance, and participant satisfaction of the intervention protocol, and processes for training and engaging a CHW for intervention delivery in preparation for a larger, fully powered trial will be assessed. Secondary aims will include health outcomes that indicate promise of the intervention's potential effect on cardiovascular risk reduction and will include measurement of hemoglobin A1c, lipid panel, blood pressure, body anthropometrics and nutritional intake (food frequency questionnaire, diet quality with HEI (healthy eating index) scoring, Veggie Meter scores as an indicator of adherence to intervention). These risk factor outcomes will be measured at baseline, 18 weeks (intermediate feasibility) and at 30 weeks to evaluate long term feasibility of the project among older adults participating in a congregate meal program.

ELIGIBILITY:
Inclusion Criteria:

* community dining site with a minimum of 20 or more congregate meal program participants.
* ≥ 60 years of age
* registered meal program participant at the community dining site
* speak English

Exclusion Criteria:

* less than 60 years of age
* don't participate in baseline measurements

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible individuals who enroll in the study | 6 months
  Feasibility will be measured by recruitment rates, the proportion of eligible individuals who enroll during the time required to reach enrollment targets.
Number of participants enrolled at each timepoint | Baseline, week 18, and week 30
  Retention rates at each time point will be quantified
Change in Veggie Meter scores | Baseline, week 18, and week 30
  The participant's adherence to the intervention will be assessed using the veggie meter, which uses light reflectance spectroscopy to provide an estimated skin carotenoid composite score. Score ranges from 0 to 800, with higher scores associated with greater fruit and vegetable intake.
Participant Satisfaction with intervention | 30 weeks
  Overall satisfaction will be measured using a likert type scale 0-5, with a higher score equating to greater satisfaction, satisfaction will include measurement of frequency, duration and timing of intervention, total scores will range from 0-15, a mean score for overall satisfaction will be reported

SECONDARY OUTCOMES:
Change in hemoglobin A1c | baseline, 18 weeks and 30 weeks
  Hemoglobin A1c will be measured with the Bayer HgA1c point of care machine
Change in total cholesterol per lipid panel | Baseline, 18 and 30 weeks
  Lipids will be measured using Cholestech LDX point of care machine using fingerstick non-fasting blood samples,
Change in systolic blood pressure | baseline, 18 and 30 weeks
  Measurement of systolic blood pressure will be obtained using a digital BP machine
Change in diastolic blood pressure | baseline, 18 and 30 weeks
  Measurement of diastolic blood pressure will be obtained using a digital BP machine
Change in waist circumference | baseline, 18 and 30 weeks
  Waist circumference will be measured using a cloth measuring tape at the point of the umbilicus with minimal clothing
Change in diet quality using an HEI index score | baseline, 18 and 30 weeks
  Diet quality will be assessed using a Frequency Questionnaire (FFQ). The NDSR FFQ provides the data that allows for calculating the Healthy Eating Index. We will use the 2015 index rules. Healthy Eating Index (HEI) 2015 Score and individual component scores will be calculated from the FFQ according to the HEI-2015 guidelines to assess changes in overall diet quality and changes within each component. The range of scores for the Healthy Eating Index 2015 is 0-100. A higher score is considered better and represents meeting more of the recommended dietary guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Martha Biddle, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No